CLINICAL TRIAL: NCT06688825
Title: Feasibility Study for the Comprehensive Overweight/Obesity Management Pre-Kidney Transplant (COMPKT) Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Society of Health-System Pharmacists Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20029799
Record Dates: First submitted 2024-10-29; First posted 2024-11-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant; Complications; Obesity
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This project will be a single-arm feasibility study, with a treatment intervention that includes three interrelated components: (1) patient education using a proven weight loss curriculum, and (2) technology tools for making healthy lifestyle choices.
Masking Description: This project will be a single-arm feasibility study, with a treatment intervention that includes three interrelated components: (1) patient education using a proven weight loss curriculum, and (2) technology tools for making healthy lifestyle choices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects on the waiting list for kidney transplant at VCUHS with BMI greater than 35 kg/m2. (Experimental): This project will be a single-arm feasibility study, with a treatment intervention that includes three interrelated components: (1) the use of medications for weight loss, (2) patient education using a proven weight loss curriculum, and (3) technology tools for making healthy lifestyle choices.
  Interventions: Behavioral: Education regarding Weight loss; Behavioral: Lifestyle tools for weight loss; Biological: Blood draw

INTERVENTIONS:
Behavioral: Education regarding Weight loss — Per American Association of Clinical Endocrinology (AACE) guidelines
Behavioral: Lifestyle tools for weight loss — Calorie App, Continuous GlucosWe Monitor (CGM), Weight Scale, Food Scale
Biological: Blood draw — Per American Association of Clinical Endocrinology (AACE) guidelines

SUMMARY:
This project will be a single-arm feasibility study, with a treatment intervention that includes three interrelated components: (1) patient education using a proven weight loss curriculum, and (2) technology tools for making healthy lifestyle choices.

DETAILED DESCRIPTION:
To optimize care for overweight/obese patients who are awaiting kidney transplants by implementing a referral process and a multi-pronged, team-based nurse/pharmacist/dietitian weight loss treatment intervention to help these patients achieve transplant criteria. Obesity, hypertension, and ESRD disproportionately affect the Black community, and Black patients have been historically disadvantaged by race-inclusive calculations that overestimated their kidney function. Effective January 5, 2023, the Organ Procurement and Transplantation Network Board of Directors requires use of a race-neutral estimated glomerular filtration rate (eGFR) to qualify candidates for kidney transplant. They also required transplant programs to identify Black candidates who may have been wrongly denied qualification

ELIGIBILITY:
Inclusion Criteria:

* on the waiting list for kidney transplant at VCUHS
* BMI greater than 35 kg/m2

Exclusion Criteria:

* Children, prisoners, pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life-Lite survey | Only completed at baseline and week 40
  Impact of Weight on Quality of Life-Lite (IWQOL-Lite©) Screening. IWQOL-Lite© is a validated, 31-item, self-report measure of obesity-specific quality of life in adults. The scale structure of the IWQOL-Lite has been verified with confirmatory factor analysis.
  In addition to a total score, there are scores on five domains:
  Physical function (11 items) Self-esteem (7 items) Sexual life (4 items) Public distress (5 items) Work (4 items)
  Scores range from 0 to 100, with 100 representing the best quality of life.
Meal recall survey | completed at weeks 1, 4, 8, 12, 20 and 28
  A meal recall survey, also known as a 24-hour dietary recall, is a structured interview that asks a person to recall what they ate and drank in the previous 24 hours. The goal is to gather detailed information about a person's diet, including portion sizes, cooking methods, and time of consumption. This information can be used to identify dietary patterns, assess nutrient intake, and develop nutrition recommendations
PrevenT2 education T | Weekly for weeks 1-12, then monthly on weeks 16, 24, 28, 32 and 36
  A program from the National Diabetes Prevention Program that helps people with prediabetes to change their risk of developing type 2 diabetes using a CDC-approved curriculum. The PreventT2 program can help people with prediabetes cut their risk of developing type 2 diabetes in half. T

CONTACTS AND LOCATIONS:
Overall Officials: Evan Sisson, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States